CLINICAL TRIAL: NCT05612737
Title: Histological and Raman Spectroscopy Evaluation of Edentulous Alveolar Ridge Horizontal Bone Augmentations Using a Xenogeneic Bone Substitute and Autologous Platelet Concentrates: A Prospective Case Series
Brief Title: Evaluation of a Novel Horizontal Ridge Augmentation Technique in Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Purgo Biologics Inc. (Unknown); FORM-Lab (Unknown)
Responsible Party: Principal Investigator, Pal Nagy, Assistant Professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HORAUG
Record Dates: First submitted 2022-10-30; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Bone Augmentation; Bone Loss, Alveolar
Keywords: platelet concentrate; horizontal bone augmentation; "sticky bone"; Histology; Raman spectroscopy
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: All subjects undergo the same type of horizontal bone augmentation using "sticky bone" (combination of xenograft and autologous platelet rich concentrate) and tenting screws.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Sticky bone" and tenting screw (Experimental)
  Interventions: Procedure: Horizontal bone augmentation

INTERVENTIONS:
Procedure: Horizontal bone augmentation — After taking six 9 mL tubes of blood from the patient, advanced (A-PRF) and liquid (S-PRF) PRFs were prepared. A-PRF was chopped, added to the xenogeneic bone substitute (THE Graft; Purgo Biologics Inc.), and then impregnated with the liquid S-PRF, which enabled the particulate bone substitute to become moldable and turned into a block ("sticky bone"). After local anesthesia, a midcrestal incision was made with one vertical releasing incision at the flap's mesial end. After full-thickness flap elevation, a periosteal releasing incision was made at the flap's apical portion. The alveolar bone was decorticalized on the buccal aspect with surgical burs. Next, the prepared "bonded" graft matrix was adapted to the ridge. Then, tenting screws (Pro-fix; Osteogenics) were placed to maintain the periosteum in an elevated and tension-free position The bone augmentation material was covered with A-PRF membranes. Finally, tension-free wound closure was performed.

SUMMARY:
This case series aimed to assess the efficacy of a novel horizontal ridge augmentation modality using histomorphometry and Raman spectroscopy. Combinations of "sticky bone" and tenting screws without autologous bone were used as augmentative materials.

DETAILED DESCRIPTION:
This case series aimed to evaluate the efficacy of the horizontal augmentation technique using the tenting screw technique with "sticky bone." The main aim was to determine whether this method provides similar results to the gold standard GBR or autologous onlay block grafts. In addition, the validity of neglecting autologous graft and its possible substitution with growth factor concentrate were examined. The novelty of this study is that no human histological examination of the described procedure has been conducted previously. It is hypothesized that the "stick bone" containing autologous platelet concentrate can substitute the use of particulate autologous bone graft in these type of procedures. In this prospective case series study five patients were enrolled and treated with the same type of bone augmentation in order to increase the alveolar ridge in the horizontal dimension with the previously mentioned technique. After 5 months of healing a second reentry surgery was performed in order to harvest the bone core for biopsy, to asses the chemical compound composition by Raman spectroscopy in vivo and to place the dental implants at the same time. Newly formed tissues were evaluated clinically during reentry, radiologically by CBCT acquisition, qualitatively and quantitatively by histological processing and physicochemically by means of Raman spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* one or more missing teeth in the jaw's posterior area, where horizontal bone width is ≤5 mm.
* no deficiency in the vertical dimension.
* The tooth must have been removed ≥4 months before augmentation.
* The patient should understand the nature of the research and be compliant in study-related activities

Exclusion Criteria:

* pregnancy
* smoking
* uncontrolled diabetes
* systemic diseases or drug consumption affecting bone metabolism, and clinically relevant osteoporosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Amount of newly formed bone by means of histomorphometry | 5 months postoperatively
  The percentage of newly formed bone of the augmented site within the biopsy
Amount of graft material bone by means of histomorphometry | 5 months postoperatively
  The percentage of graft material (THE Graft; Purgo Biologics Inc.) of the augmented site within the biopsy
Amount of soft tissue by means of histomorphometry | 5 months postoperatively
  The percentage of soft tissue of the augmented site within the biopsy
The quality of the newly formed tissues by means of histology | 5 months postoperatively
  The descriptive analyses of the cells and tissue structure of the augmented site within the biopsy

SECONDARY OUTCOMES:
In vivo spectroscopy analyses of the augmented site with a Raman spectrometer device | 5 months postoperatively
  Raman investigation (measuring wavelength in the range 300-1800 cm-1) highlights the peaks (Raman shift) for the main bone components (chemical groups and elements) in order to evaluate differences between bone tissue for the investigated patients. Differences in peaks intensity on raw spectra reflected the differences in the quantities of the chemical components for investigated specimens.
CBCT analysis | 5 months postoperatively
  Horizontal bone volume gain (measured in mm) evaluated on pre- and postoperative CBCT-s.
The clinical descriptive bone assessment of the augmented bone site | 5 months postoperatively
  The descriptive clinical assessment is a subjective evaluation of the augmented bone judged by the operator. The presence of possibly occuring non-integrated graft remnants can be assessed during reentry surgery.
The clinical descriptive bone assessment of the augmented bone site | 5 months postoperatively
  The descriptive clinical assessment is a subjective evaluation of the augmented bone judged by the operator. The bleeding property of the newly formed bone after drilling the osteotomy for the implant can be assessed during reentry.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urban IA, Nagursky H, Lozada JL, Nagy K. Horizontal ridge augmentation with a collagen membrane and a combination of particulated autogenous bone and anorganic bovine bone-derived mineral: a prospective case series in 25 patients. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):299-307. doi: 10.11607/prd.1407. PMID 23593623
- [Background] Khoury F, Hanser T. Mandibular bone block harvesting from the retromolar region: a 10-year prospective clinical study. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):688-97. doi: 10.11607/jomi.4117. PMID 26009921
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Farias D, Caceres F, Sanz A, Olate S. Horizontal Bone Augmentation in the Posterior Atrophic Mandible and Dental Implant Stability Using the Tenting Screw Technique. Int J Periodontics Restorative Dent. 2021 Jul-Aug;41(4):e147-e155. doi: 10.11607/prd.5137. PMID 34328475
- [Background] Gheno E, Alves GG, Ghiretti R, Mello-Machado RC, Signore A, Lourenco ES, Leite PEC, Mourao CFAB, Sohn DS, Calasans-Maia MD. "Sticky Bone" Preparation Device: A Pilot Study on the Release of Cytokines and Growth Factors. Materials (Basel). 2022 Feb 16;15(4):1474. doi: 10.3390/ma15041474. PMID 35208017
- [Background] Ghanaati S, Booms P, Orlowska A, Kubesch A, Lorenz J, Rutkowski J, Landes C, Sader R, Kirkpatrick C, Choukroun J. Advanced platelet-rich fibrin: a new concept for cell-based tissue engineering by means of inflammatory cells. J Oral Implantol. 2014 Dec;40(6):679-89. doi: 10.1563/aaid-joi-D-14-00138. PMID 24945603